CLINICAL TRIAL: NCT03080272
Title: The Goal of "no Worse Than Mild Pain" in Daily Clinical Practice: Individual Responder Analysis - a Cross-sectional Prospective Cohort Study of Surgical Patients at Zealand University Hospital, Koege
Brief Title: Do we Achieve the Goal of "No Worse Than Mild Pain" in Daily Clinical Practice?
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Anja Geisler, Clinical nurse specialist / PhD student, Zealand University Hospital
Other Study IDs: SM3-AG-2017
Record Dates: First submitted 2017-02-27; First posted 2017-03-15 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Pain, Postoperative
Keywords: individual patient
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Spinal Surgery: No intervention will take place. Recruiting Autumn 2017 until spring 2018
  Interventions: Other: no intervention will take place
- Gastric sleeve: No intervention will take place. Recruiting Autumn 2017 until spring 2018
  Interventions: Other: no intervention will take place
- Total knee arthroplasty: No intervention will take place. Recruiting Spring 2018 until Summer 2018
  Interventions: Other: no intervention will take place
- Shoulder arthroplasty: No intervention will take place. Recruiting Winter 2017 until Summer 2018
  Interventions: Other: no intervention will take place
- Maxillofacial surgery: No intervention will take place. Recruiting 6 march 2017 until Autumn 2017
  Interventions: Other: no intervention will take place

INTERVENTIONS:
Other: no intervention will take place — Only registration and data collection of patients' care and treatment will take place. There will be no changes in patients' treatment. No intervention will take place

SUMMARY:
With this study the investigators want to perform a prospective cross-sectional audit at Zealand University Hospital, Koege, Denmark. The aim is to investigate the actual pain treatment and outcomes from a representative number of surgical procedures from different surgical departments.

DETAILED DESCRIPTION:
In contemporary postoperative pain management, patients are treated with combinations of non-opioid and opioid analgesics, and analgesic methods. The intention is to enhance pain relief from additive or synergistic effects of such combinations. However, the literature is complex and heterogenic and characterized by small sized studies investigating a diversity of analgesic combinations and methods. Consequently no well-documented "best current proven intervention" is definable

Efficacy of analgesics is most often based on results from randomized trials measuring differences between two groups based on the average pain level in each group, for example median or mean. This approach has weaknesses as individual patients vary in response, and the average pain level is actually only experienced by few patients. Also, it is well known that analgesics may only work in 30- 50% of the patients and it is not possible to predict who will experience excessive pain. Besides, data on pain score does not follow a normal distribution, but usually is either very good or very bad. Studies have demonstrated, that basically, patients want efficient pain treatment with large pain reductions (for example 50%) and/or pain levels corresponding to mild pain, Numeric Rating Scale ≤ 3. Pain treatment that does not include the achievement of adequate pain relief are likely to fail.

Consequently, a new and simple universal criterion for postoperative analgesic success has been suggested based on individual patient response analyses: Efficacy should be measured on the individual level, and patients should experience "no worse than mild pain"(Numeric Rating Scale ≤ 3). In a re-calculation of individual patient data from 16 randomized clinical trials, the investigators have recently documented that by using the success criteria that at least 80% of patients should achieve Visual Analogue Scale ≤ 30, only about 50% of the studies had achieved goal fulfillment.

A current review has further documented, that movement evoked pain is underreported. Only 39% of trials measured movement evoked pain even though trials measuring both movement evoked pain and pain at rest suggest that movement evoked pain is 95% - 226% more severe and intense for the patient than pain at rest. Therefore it is of great importance for the benefits and treatment of patients, that future trials not only record pain at rest but also movement evoked pain, and additionally supply relevant information about the actual physical maneuver used for assessment.

It is therefore essential, in the light of "no worse than mild pain", and based on individual responder analysis, to investigate current benefit and harm of postoperative pain treatment. Our goal is to highlight the need for an intensified focus on individual patient's pain and the investigators expect to shed a new and critical light on current clinical pain treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following criteria to be suitable for inclusion in the study

* Age > 18 år
* Patients scheduled for relevant surgical procedure
* Patients who understand and speak Danish or English -

Exclusion Criteria:

Patients who meet one or more of the following criteria are not suitable for inclusion in this study:

* Patients who cannot cooperate
* Alcohol and drug dependency as judged by the investigator
* Chronic opioid dependent patients

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a relevant surgical intervention at Zealand University Hospital, Koege and meeting the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Pain during mobilisation late | Outcome measure will be assessed and data will be presented in june 2018
  Proportions achieving "no worse than mild pain" (Numeric Rating Scale ≤ 3) for pain during mobilisation at 24 hours (±2h) postoperatively

SECONDARY OUTCOMES:
Pain during mobilisation early | Outcome measure will be assessed and data will be presented in june 2018
  Proportions achieving "no worse than mild pain" (Numeric Rating Scale ≤ 3) during mobilisation at 6 hours (±2h) postoperatively
Pain at rest early | Outcome measure will be assessed and data will be presented in june 2018
  Proportions achieving "no worse than mild pain" (Numeric Rating Scale ≤ 3) at rest at 6h (±2h) and 24h (±2h) postoperatively
Numeric Rating Scale pain levels | Outcome measure will be assessed and data will be presented in june 2018
  Numeric Rating Scale pain levels at rest and during mobilisation at 6h (±2h) and 24h (±2h) after completed surgery 6 and 24 hours
Patient satisfaction | Outcome measure will be assessed and data will be presented in june 2018
  Patients' experience of pain treatment and their contentment hereof using a questionnaire based on "PAIN OUT" at 24h (±2h) postoperatively
Morphine consumption | Outcome measure will be assessed and data will be presented in june 2018
  Morphine i.v. equivalent consumption (mg) the first 24h postoperatively (including opioids given as pre-medication
Non opioid use | Outcome measure will be assessed and data will be presented in june 2018
  Non-opioid analgesic usage the first 24h postoperatively (including non-opioids given as pre-medication)
Nausea | Outcome measure will be assessed and data will be presented in june 2018
  Nausea measured by Verbal Rating Scale at T6 og T24 hours postoperatively
Vomiting | Outcome measure will be assessed and data will be presented in june 2018
  Vomiting (number of episodes 0-24 hours) postoperatively
Dizziness | Outcome measure will be assessed and data will be presented in june 2018
  Dizziness measured by Verbal Rating Scale at T6 and T24 hours
Sedation | Outcome measure will be assessed and data will be presented in june 2018
  Sedation measured by Verbal Rating Scale at T6 og T24 hours postoperatively
LOS | Outcome measure will be assessed and data will be presented in june 2018
  Length of postoperative hospital stay measured in days
Readmission | Outcome measure will be assessed and data will be presented in june 2018
  Re-admission within 90 days postoperatively
Mortality | Outcome measure will be assessed and data will be presented in june 2018
  Mortality within the first 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Ole Mathiesen, MD.PhD, Study Director — Zealand University Hospital, Koege
Locations (1):
- Zealand University Hospital, Køge, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
no plan

REFERENCES:
- [Background] Kehlet H. Fast-track surgery-an update on physiological care principles to enhance recovery. Langenbecks Arch Surg. 2011 Jun;396(5):585-90. doi: 10.1007/s00423-011-0790-y. Epub 2011 Apr 6. PMID 21468643
- [Background] Kehlet H, Dahl JB. Anaesthesia, surgery, and challenges in postoperative recovery. Lancet. 2003 Dec 6;362(9399):1921-8. doi: 10.1016/S0140-6736(03)14966-5. PMID 14667752
- [Background] Dahl JB, Mathiesen O, Kehlet H. An expert opinion on postoperative pain management, with special reference to new developments. Expert Opin Pharmacother. 2010 Oct;11(15):2459-70. doi: 10.1517/14656566.2010.499124. PMID 20586709
- [Background] Rathmell JP, Wu CL, Sinatra RS, Ballantyne JC, Ginsberg B, Gordon DB, Liu SS, Perkins FM, Reuben SS, Rosenquist RW, Viscusi ER. Acute post-surgical pain management: a critical appraisal of current practice, December 2-4, 2005. Reg Anesth Pain Med. 2006 Jul-Aug;31(4 Suppl 1):1-42. doi: 10.1016/j.rapm.2006.05.002. PMID 16849098
- [Background] Gurusamy KS, Vaughan J, Toon CD, Davidson BR. Pharmacological interventions for prevention or treatment of postoperative pain in people undergoing laparoscopic cholecystectomy. Cochrane Database Syst Rev. 2014 Mar 28;2014(3):CD008261. doi: 10.1002/14651858.CD008261.pub2. PMID 24683057
- [Background] Hojer Karlsen AP, Geisler A, Petersen PL, Mathiesen O, Dahl JB. Postoperative pain treatment after total hip arthroplasty: a systematic review. Pain. 2015 Jan;156(1):8-30. doi: 10.1016/j.pain.0000000000000003. PMID 25599296
- [Background] Moore A, Derry S, Eccleston C, Kalso E. Expect analgesic failure; pursue analgesic success. BMJ. 2013 May 3;346:f2690. doi: 10.1136/bmj.f2690. No abstract available. PMID 23645858
- [Background] Moore RA, Straube S, Aldington D. Pain measures and cut-offs - 'no worse than mild pain' as a simple, universal outcome. Anaesthesia. 2013 Apr;68(4):400-12. doi: 10.1111/anae.12148. Epub 2013 Jan 24. No abstract available. PMID 23347230
- [Background] Geisler A, Dahl JB, Karlsen AP, Persson E, Mathiesen O. Low degree of satisfactory individual pain relief in post-operative pain trials. Acta Anaesthesiol Scand. 2017 Jan;61(1):83-90. doi: 10.1111/aas.12815. Epub 2016 Oct 3. PMID 27696343
- [Background] Srikandarajah S, Gilron I. Systematic review of movement-evoked pain versus pain at rest in postsurgical clinical trials and meta-analyses: a fundamental distinction requiring standardized measurement. Pain. 2011 Aug;152(8):1734-1739. doi: 10.1016/j.pain.2011.02.008. Epub 2011 Mar 12. PMID 21402445
- [Derived] Geisler A, Zachodnik J, Nersesjan M, Persson E, Mathiesen O. Postoperative Pain Management and Patient Evaluations After Five Different Surgical Procedures. A Prospective Cohort Study. Pain Manag Nurs. 2022 Dec;23(6):791-799. doi: 10.1016/j.pmn.2022.06.006. Epub 2022 Aug 6. PMID 35941015